CLINICAL TRIAL: NCT03962231
Title: Rotator Cuff Unloading Versus Loading Exercise Program in Patients With Shoulder Pain and Rotator Cuff Tear: a Randomized Clinical Trial
Brief Title: Exercise Program in Patients With Shoulder Pain and Rotator Cuff Tear
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Larissa Pechincha Ribeiro (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor-Investigator, Larissa Pechincha Ribeiro, Principal Investigator, Universidade Federal de Sao Carlos
Organization: Universidade Federal de Sao Carlos (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UFSCarShoulderLabRC
Record Dates: First submitted 2019-05-20; First posted 2019-05-23 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Shoulder Pain; Rotator Cuff Injuries; Rehabilitation
Keywords: Treatment; Physiotherapy; Impingement Syndrome
MeSH Terms: conditions — Shoulder Pain; Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rotator Cuff Unloading Exercise Program (Active Comparator): Patients in this group will perform semi-closed kinetic chain elevation exercises, deltoid re-education exercises, assisted arm elevation and scapula control exercises.
  Interventions: Other: Rotator Cuff Unloading Exercise Program
- Rotator Cuff Loading Exercise Program (Active Comparator): Patients in this group will perform conventional exercises with focus on lateral rotation, medial rotation and arm elevation.
  Interventions: Other: Rotator Cuff Loading Exercise Program

INTERVENTIONS:
Other: Rotator Cuff Unloading Exercise Program — Patients in this group will perform semi-closed kinetic chain elevation exercises, deltoid reeducation exercises, assisted arm elevation and scapular control exercises.
  Arms: Rotator Cuff Unloading Exercise Program
Other: Rotator Cuff Loading Exercise Program — Patients in this group will perform conventional exercises focusing on lateral rotation, medial rotation and arm elevation.
  Arms: Rotator Cuff Loading Exercise Program

SUMMARY:
Introduction: Atraumatic and degenerative rotator cuff tears are common in individuals over 55 years of age. This condition can have a high impact on social life and is associated with chronic pain, weakness and dysfunction of the upper limb. There is evidence that conservative approaches should be the first treatment option. Conservative treatment usually addresses a variety of therapeutic behaviors without providing scientific arguments for the choice and progression of exercises. At that, there is a gap in the literature on the best exercises for this population, whether they are exercises to strengthen the remaining fibers of the rotator cuff or exercises focused on strengthening other shoulder muscles with rotator cuff unload exercise program. Objective: To compare the effects of two different exercise programs based on the load of the rotator cuff on a population with shoulder pain and rotator cuff tear. Methods: This is a controlled, randomized, blinded clinical trial. In this study 78 individuals with shoulder pain and presence of atraumatic rupture of the rotator cuff muscle tendon will participate and will be randomly distributed between two groups. The primary outcome will be quality of life (WORC index), and secondary outcomes will include pain, function (DASH), fear avoidance beliefs (FABQ-Brazil), kinesiophobia (Tampa Scale), pain catastrophizing scale, muscle strength of abductors, lateral and medial rotators of the shoulder, range of motion of arm elevation and patient satisfaction. All outcomes will be measured before and after 12 weeks of treatment (2x/week), and 1 month after the end of treatment. The normality of the data will be verified by the Kolmogorov Smirnov test. The differences between the groups will be verified using the mixed linear models with the terms of interaction versus time. The effect size will be calculated for the variables between the groups. The level of significance will be 5%.

DETAILED DESCRIPTION:
BACKGROUND The presence of atraumatic and degenerative ruptures in the rotator cuff is a common finding in imaging studies due to the natural aging process. Several exercise protocols have been proposed for this population. However, there is still a gap in the literature about what exercises are best for these individuals: exercises to strengthen the remaining fibers of the rotator cuff or exercises focused on strengthening other shoulder muscles with little emphasis on the rotator cuff. Both types of exercises are performed jointly in most treatment programs, or the tension in the rotator cuff is not taken into account during exercise selection.

Despite the lack of consensus on which exercises or exercises are more effective in conservative treatment, there is evidence that therapeutic exercises should be the first treatment option in individuals with chronic, atraumatic, degenerative, and rotator cuff tears. Thus, it is expected that this study may contribute to filling the existing gap, re-adjusting treatment techniques for this population and provide scientific bases that support the clinical practice of physiotherapists.

RESEARCH QUESTION:

Are the results of a rotator cuff unloading exercise program different than rotator cuff loading exercise program in individuals with shoulder pain and rotator cuff tear? This research question is relevant to clinical practice once that so far there are no specific treatment guidelines for patients with degenerative ruptures of the rotator cuff tendons.

Primary Aim The primary aim of this study will be to verify the effects of 12-week unloading rotator cuff exercise program compared to an usual exercise program with an emphasis on the rotator cuff on quality of life in patients with shoulder pain and and rotator cuff tear.

Secondary Aim

The secondary aim will be to verify the effects of 12-week unloading rotator cuff exercise program compared to an usual exercise program with an emphasis on the rotator cuff on quality of life in patients with shoulder pain and and rotator cuff tear following variables:

* Pain at rest, during arm movement, maximum and minimum referred in the last week;
* Function of upper limbs;
* Fear-Avoidance Beliefs;
* Kinesiophobia;
* Pain Catastrophizing;
* Strength of abductors, lateral and medial rotators of the shoulder;
* Range of movement during arm elevation;
* Satisfaction of patients with the treatment;

HYPOTHESES The hypothesis of this study is that the exercise program with no emphasis on the rotator cuff will produce different results on quality of life, pain, function, fear-avoidance beliefs, kinesiophobia, pain catastrophizing, muscle strength of abductors, lateral and medial rotators of the arm, range of motion during arm elevation and treatment satisfaction when compared to the exercise program with an emphasis on the rotator cuff.

METHODOLOGY

1. Study Design Controlled, randomized, blind and two-group clinical trial parallel. Evaluators will be blinded to the treatment group.
2. Ethical Aspects This study was sent to the Research Ethics Committee of the University and registered in clinicaltrials.gov, respecting the norms of experimental conduct with humans (CNS Resolution 466/12). Participants will receive verbal and written explanation of the research objectives and procedures. They will also be informed of all the risks and benefits of their participation, as well as the freedom to give up participating in the research at any time. Individuals who agree to participate will sign the Free and Informed Consent Form. Any changes that are made to the research protocol will be submitted to the UFSCar Research Ethics Committee and registered at clinicaltrials.gov.
3. Sample The sample size was performed based on the minimum important difference of 282.6 points of the Western Ontario Rotator Cuff Index (WORC) 50 with standard deviation of 400 points, 80% power, and significance level of 5%. WORC was selected because it evaluates the quality of life of individuals with rotator cuff diseases. Considering a sample loss of 15%, 9 will be included in the study 78 subjects, randomly assigned to two treatment groups: Rotator Cuff Unloading Exercise Program (n = 39) and Rotator Cuff Loading Exercise Program (n = 39).

Block randomization between groups will be performed by the site www.randomization.com and the sequence will be stored in sealed and opaque envelopes to maintain allocation secrecy. This process will be performed by an independent researcher, that is, who will not be involved with the evaluation and treatment. The allocation of individuals will be revealed to the investigator responsible for the treatment with the opening of the envelope before the beginning of the intervention. The researcher responsible for the evaluation will be blinded on the treatment group. The subjects will be blinded to the hypothesis of the study, and in addition, the treatment will be performed individually, that is, they will not have contact between the participants of the same or the other group.

STATISTICAL ANALYSIS Recruitment information and data of subjects included, and dropouts of all evaluations will be collected and manually inserted into Excel software (Microsoft version 2016). The confidentiality of the data will be guaranteed by transforming the individuals' names into identifier codes. In addition, only study researchers will have access to survey material and database.

Statistical Package for Social Sciences version 23 will be used to analyze the data. Continuous data will be presented by mean, standard deviation and mean difference between the groups with 95% confidence interval, and the categorical ones by frequency and percentage. The normality of the data will be verified through the Kolmogorov Smirnov test and observation of histograms for each variable in each group. Statistical analysis will follow the principles of intention-to-treat analysis.

Linear mixed models will be used to calculate the differences between the groups using the terms of group interaction (Rotator Cuff Unloading Exercise Program and Rotator Cuff Loading Exercise Program) versus time (pre-treatment, 12 weeks at the end of treatment, and one month after the end of treatment) for the variables of quality of life (WORC index), pain, function (DASH questionnaire), fear-avoidance beliefs (FABQBrasil), kinesiophobia, pain catastrophizing scale (PCS), muscle strength of abductors, lateral and medial rotators of the shoulder and range of motion of arm elevation. The models will be adjusted to baseline values for all variables and for multiple comparisons.

The effect size will also be calculated between groups, where an effect greater than 0.8 will be considered large, about 0.5 moderate, and less than 0.2 small.80 A significance level of 5% (p <0.05).

ELIGIBILITY:
Inclusion Criteria:

* age 55 years or over;
* shoulder pain;
* at least 90° of arm elevation;
* atraumatic rotator cuff tear.

Exclusion Criteria:

* Individuals with a history of trauma associated with onset of symptoms;
* fracture and/or previous surgery on upper limbs;
* pain related to the cervical spine;
* inflammatory arthritis;
* adhesive capsulitis;
* cognitive alteration that makes it impossible to perform the questionnaires.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2019-08-05 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Quality of Life at 12 weeks and 1 month (follow-up) - The Western Ontario Rotator Cuff Index (WORC) | Pre (baseline) treatment, post treatment (12 weeks) and after 1 month (follow-up)
  The Western Ontario Rotator Cuff Index (WORC) contains 21 questions distributed in five domains, each question can be scored between 0 and 100 on the Analogic visual scale. The final result of WORC varies from 0 to 2100, higher value indicates worse the quality of life of the individual.

SECONDARY OUTCOMES:
Change from Baseline Shoulder Pain at 12 weeks and 1 month (follow-up) | Pre (baseline) treatment, post treatment (12 weeks) and after 1 month (follow-up)
  The pain will be measured with 11 point - Numerical Rating Pain Scale with scores ranging from 0 (no pain) to 10 (maximum pain).
Change from Baseline Upper Limb Function at 12 weeks and 1 month (follow-up) | Pre (baseline) treatment, post treatment (12 weeks) and after 1 month (follow-up)
  The Function will be measured with Disabilities of the Arm, Shoulder and Hand with scores ranging from 0 to 100 (higher score reflects greater disability)
Change from Baseline Fear Avoidance Beliefs at 12 weeks and 1 month (follow-up) | Pre (baseline) treatment, post treatment (12 weeks) and after 1 month (follow-up)
  The Fear-Avoidance Beliefs Questionnaire (FABQ) contains 2 scales: FABQ work scale (with range from 0 to 42) and FABQ physical activity scale (with range from 0 to 24). Higher scores indicate higher levels of fear-avoidance beliefs.
Change from Baseline Kinesiophobia at 12 weeks and 1 month (follow-up) | Pre (baseline) treatment, post treatment (12 weeks) and after 1 month (follow-up)
  The Kinesiophobia will be measured with Tampa Scale of Kinesiophobia (TKS) with scores ranging from 17 to 68. Higher scores indicate higher degree of kinesiophobia.
Change from Baseline Pain Catastrophizing at 12 weeks and 1 month (follow-up) | Pre (baseline) treatment, post treatment (12 weeks) and after 1 month (follow-up)
  The Pain Catastrophizing Scale is self-administered and contains 13 items. Scale scores range from 0 to 52, with higher values indicating a higher degree of catastrophic thoughts.
Change from Baseline Muscle Strength at 12 weeks and 1 month (follow-up) | Pre (baseline) treatment, post treatment (12 weeks) and after 1 month (follow-up)
  The abductors, lateral and medial rotators of the arm will be tested using handheld dynamometer.
Change from Baseline Range of Motion at 12 weeks and 1 month (follow-up) | Pre (baseline) treatment, post treatment (12 weeks) and after 1 month (follow-up)
  The maximum range of motion during arm elevation, the range of onset and end of pain in the sagittal and scapular planes will be recorded using a digital inclinometer.
Change from Baseline self-perception of improvement at 12 weeks and 1 month (follow-up) | Post treatment (12 weeks) and after 1 month (follow-up)
  The Overall improvement of Symptoms will be measured with the Global Rating of Change Scale with scores ranging from -7 to +7 (A higher score indicates higher recovery from the condition).

CONTACTS AND LOCATIONS:
Overall Officials: Larissa P Ribeiro, MD, Principal Investigator — Department of Physical Therapy - Universidade Federal de São Carlos
Locations (1):
- Federal University of Sao Carlos, São Carlos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
At the end of the clinical trial will be published the Study Protocol and Statistical Analysis Plan (SAP), if any researcher wants more information can request. The Informed Consent Form (ICF) can also be available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: at the end of the study
Access Criteria: At the end of the clinical trial will be published the Study Protocol and Statistical Analysis Plan (SAP), if any researcher wants more information can request. The Informed Consent Form (ICF) can also be available. Any researcher can request more information.

REFERENCES:
- [Derived] Ribeiro LP, Cools A, Camargo PR. Rotator cuff unloading versus loading exercise program in the conservative treatment of patients with rotator cuff tear: protocol of a randomised controlled trial. BMJ Open. 2020 Dec 12;10(12):e040820. doi: 10.1136/bmjopen-2020-040820. PMID 33310803